CLINICAL TRIAL: NCT01346683
Title: An Open, Prospective, Multi-center Study to Evaluate the OsseoSpeed™ TX Implant With an Early Loading Protocol in Patients With Tooth Loss in the Posterior Mandible. A 3-years Follow-up Study.
Brief Title: Study on OsseoSpeed™ TX Implants in a Chinese Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-0002
Record Dates: First submitted 2011-05-02; First posted 2011-05-03 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Partially Edentulous Jaw
MeSH Terms: conditions — Jaw, Edentulous, Partially

ARMS (1):
- OsseoSpeed TX (Experimental): OsseoSpeed TX implants of lengths 8-17 mm
  Interventions: Device: OsseoSpeed TX

INTERVENTIONS:
Device: OsseoSpeed TX — OsseoSpeed TX implants of lengths 8-17 mm

SUMMARY:
To investigate the clinical efficacy of OsseoSpeed™ TX implants in a Chinese population by evaluation of marginal bone level alteration, implant stability and implant survival in the posterior mandible up to 3 years after loading. Hypothesis: Early loading of the posterior mandible is a safe and predictable procedure.

ELIGIBILITY:
Inclusion criteria:

1. Provision of informed consent
2. Aged 20-75 years at enrolment
3. History of edentulism in the posterior mandible, Kennedy classes I or II, of at least four months. Last natural tooth in function is canine or first bicuspid.
4. Neighboring tooth to the planned bridge must have natural root.
5. Presence of natural teeth, partial prosthesis and/or implants in the opposite jaw in contact with the planned bridge.
6. Deemed by the investigator to have adequate bone height and a bone width of minimum 5.5 mm.
7. Deemed by the investigator as likely to present an initially stable implant situation

Exclusion criteria:

1. Unlikely to be able to comply with study procedures, as judged by the investigator
2. Earlier graft procedures in the study area
3. Current need for pre-surgical bone or soft tissue augmentation in the planned implant area.
4. Uncontrolled pathologic processes in the oral cavity
5. Known or suspected current malignancy
6. History of radiation therapy in the head and neck region
7. History of chemotherapy within 5 years prior to surgery
8. Systemic or local disease or condition that could compromise post-operative healing and/or osseointegration
9. Uncontrolled diabetes mellitus
10. Corticosteroids or any other medication that could influence post-operative healing and/or osseointegration
11. Smoking more than 10 cigarettes/day
12. Present alcohol and/or drug abuse
13. Involvement in the planning and conduct of the study (applies to both Astra Tech staff and staff at the study site)
14. Previous enrolment in the present study.
15. Simultaneous participation in another clinical study or participation in a clinical study during the last 6 months.
16. Subjects that are unable to give informed consent

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yongsheng Zhou, Prof, Principal Investigator — Department of Prosthodontics, School of Stomatology, Beijing University
Locations (3):
- China (3):
  - Department of Prosthodontics, School of Stomatology, Beijing University, Beijing
  - Department of Prosthodontics & Dental Materials, Guanghua School of Stomatology, Sun Yat-Sen University, Guangzhou
  - Department of Prosthodontics, College of Stomatology, Shanghai Jiao Tong University, Shanghai

REFERENCES:
- [Result] Zhou J, Huang Q, Wang X, Peng D, Li Y, Zhang L, Liu J, Zhang S, Zhao K, Jiang X, Zhou Y. Early loading of splinted implants in the posterior mandible: a prospective multicentre case series. J Clin Periodontol. 2016 Mar;43(3):298-304. doi: 10.1111/jcpe.12513. Epub 2016 Mar 1. PMID 26790007

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Implants
Period: Overall Study
Arm/Group | OsseoSpeed TX
Started | 45; 107 Implants
Completed | 45; 107 Implants
Not Completed | 0; 0 Implants

BASELINE CHARACTERISTICS:
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed TX
Number analyzed (Participants) | 45
Number analyzed (Implants) | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (10.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 19
Region of Enrollment [Number; unit: participants]
  China | 45

OUTCOME MEASURES:

1. Primary Outcome: Marginal Bone Level Alteration
Description: Marginal Bone Level determined from radiographs and expressed as the difference from a reference point on the implant to the most coronal bone-to-implant contact on the mesial and distal aspect of the implant. Marginal Bone Level expressed in millimeters at the 3 year follow-up visit compared to values obtained at delivery of permanent restoration i.e. loading (baseline).
Time Frame: Evaluated 3 years after implant loading
Population: Protocol deviations excluded, a total of 5 subjects (15 implants), resulting in a per protocol analysis population of 40 subjects (92 implants).
  In addition a total of 2 subjects (4 implants) had radiographs were not possible measure. Giving an analysis population of 38 subjects (88 implants) for the primary outcome measure.
Measure: Mean (Standard Deviation); unit: millimeter
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed TX
Number analyzed (Participants) | 38
Number analyzed (Implants) | 88
millimeter | 0.10 (0.61)

2. Secondary Outcome: Implant Survival
Description: Implant survival rate evaluated clinically and radiographically.
Time Frame: From implant placement to the follow-up 36 months after loading.
Population: Protocol deviations excluded, a total of 5 subjects (15 implants), resulting in a per protocol analysis population of 40 subjects (92 implants).
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed TX
Number analyzed (Participants) | 40
Number analyzed (Implants) | 92
Implants | 92

3. Secondary Outcome: Implant Stability
Description: Implant stability evaluated clinically/manually (recorded as stable yes/no)
Time Frame: Measured from loading of implants to the follow-up 36 months after loading.
Population: as for outcome 2
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed TX
Number analyzed (Participants) | 40
Number analyzed (Implants) | 92
Implants | 92

4. Secondary Outcome: Soft Tissue Status (PPD).
Description: Soft tissue status measured by assessment of probing pocket depth (PPD). PPD was measured at 4 different surfaces (mesial, distal, buccal and lingual) and change compared to baseline (loading) was analyzed.
  A negative value = increased pocket depth.
Time Frame: Measured from loading of implants to the follow-up 36 months after loading.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeter
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed TX
Number analyzed (Participants) | 40
Number analyzed (Implants) | 92
millimeter | -0.77 (0.95)

5. Secondary Outcome: Soft Tissue Status (BoP)
Description: Soft tissue status measured by assessment of bleeding on probing (BoP).
Time Frame: Measured from loading of implants to the follow-up 36 months after loading.
Population: as for outcome 2
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed TX
Number analyzed (Participants) | 40
Number analyzed (Implants) | 92
Implants | 30

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | OsseoSpeed TX
Serious Adverse Events (participants affected / at risk) | 1/45
Other Adverse Events (participants affected / at risk) | 3/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OsseoSpeed TX (N=45)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OsseoSpeed TX (N=45)
Common cold (Infections and infestations) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less